CLINICAL TRIAL: NCT04549181
Title: Enhancing Problem-Solving Skills in Underserved Rural Heart Failure Dyads
Brief Title: Problem-Solving for Rural Heart Failure Dyads
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Florida Blue Center for Rural Research (Unknown)
Responsible Party: Principal Investigator, Lucinda Graven, Associate Professor, Florida State University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 00001621
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-03

CONDITIONS: Heart Failure
Keywords: heart failure; dyads; rural; problem-solving; self-care
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Dyads (n = 60; 120 participants) will be trained to use a 4-step problem-solving process to collaboratively manage HF-related problems over 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase I: Qualitative (No Intervention): Rural HF dyads will participate in a one-time telephone-based semi-structured interview to explore the types of HF-related problems that rural HF dyads experience and how these problems are managed.
- Phase II: Problem-Solving for Rural HF Dyads (Experimental): The dyadic problem-solving intervention will be provided by a HF specialist nurse. The nurse will conduct the initial telehealth (virtual, telephone) session and provide dyads with an intervention booklet containing examples of common HF-related problems experienced by rural dyads and suggested management strategies tailored to the rural sociocultural context. The nurse will lead dyads in a card sorting task intended to help dyads prioritize current HF-related problems and will guide dyads in developing management strategies for the highest priority problem. Dyads will utilize these strategies until the next session at which time the nurse will guide dyads in evaluating the effectiveness of chosen strategies. The iterative process then begins again. Dyads will receive 7 follow-up telephone sessions with the nurse. In the intervention, the nurse will focus on problems related to self-care, including those specific to the rural population.
  Interventions: Behavioral: Phase II: Problem-Solving for Rural HF Dyads

INTERVENTIONS:
Behavioral: Phase II: Problem-Solving for Rural HF Dyads — Participants in the Intervention Group will be trained to use a 4-step problem-solving process based on the Theory of Social Problem-Solving (TSPS) to manage HF-related problems collaboratively over 12-weeks. The core belief of TSPS is effective problem-solving requires a positive problem orientation (i.e., viewing problems as a challenge versus a threat) and elicits rational problem-solving versus avoidance or impulsivity/carelessness. Dyadic problem-solving follows from a positive problem orientation and involves accurate problem identification, generation of appropriate potential solutions, active decision-making, and solution implementation and evaluation. The goal of this dyadic intervention is to move HF dyads toward a positive problem orientation and use of rational problem-solving strategies that support greater patient and family caregiver-contributed HF self-care.
  Arms: Phase II: Problem-Solving for Rural HF Dyads

SUMMARY:
This study will develop and test the effectiveness of a culturally-sensitive, telephone-based, tailored dyadic problem-solving intervention to improve self-care in rural heart failure (HF) dyads. The target population is rural-residing HF dyads (patient and family caregiver). Rural dyads will be recruited from the Florida State University Institute for Successful Longevity Participant Registry, outpatient HF/cardiac and rural healthcare clinics affiliated with the Tallahassee Memorial Hospital, Bond Community Health Clinic, via social medial and newspaper ads, and publicly available community sites (e.g., senior centers, post offices, grocery stores, etc.). Phase I (Arm I) will include a one-time telephone-based semi-structured interview. Dyads in Phase II (Arm II) will receive one telehealth (virtual or telephone) session, followed by 7 follow-up telephone sessions.

DETAILED DESCRIPTION:
The long-term goal of this research is to reduce morbidity and improve HF self-care by enhancing family problem-solving and collaborative care management among rural HF dyads. The initial step in meeting this goal is to develop and pilot-test a culturally-sensitive, telephone-based, tailored dyadic problem-solving intervention to improve HF self-care in rural HF dyads. Using a multi-phase, sequential qualitative and quantitative approach, the following research aims are to: 1) identify the major dyadic HF-related problems dyads experience and how these problems are managed; 2) develop a telephone-based, tailored dyadic problem-solving intervention and determine its feasibility and acceptability for managing HF-related problems; and 3) evaluate the preliminary effects of the telephone-based, tailored dyadic problem-solving intervention on dyadic problem-solving and patient and family caregiver contributions to HF self-care. As an exploratory aim, we will also evaluate the effectiveness of the dyadic problem-solving intervention on caregiver burden, self-care, and life changes. In Phase I, qualitative inquiry will guide in-depth semi-structured dyad interviews (n = 12-20 dyads; 24-40 participants) to identify the dyadic HF-related problems experienced by rural HF dyads and associated management strategies (Aim 1). Phase II will be guided by qualitative and quantitative methods and include a repeated measures, single-group design to evaluate the feasibility, acceptability, and preliminary effectiveness of the 12-week dyadic problem-solving intervention in a sample of rural HF dyads (n = 60 dyads; 120 participants) (Aims 2, 3). Participants for this study will be recruited from from the Florida State University Institute for Successful Longevity Participant Registry, outpatient HF/cardiac and rural healthcare clinics affiliated with Tallahassee Memorial Hospital, Bond Community Health Clinic, via social medial and newspaper ads, and publicly available community sites (e.g., senior centers, post offices, grocery stores, etc.).

Phase I (Arm 1) will identify dyadic HF-related problems and management strategies using semi-structured interviews in a sample of rural-residing HF dyads (n = 12-20 dyads; 24-40 participants). Following consent, interviews will occur once and be approximately 45 minutes long. Qualitative data from Phase I will be analyzed using thematic analytic methods and NVivo11. Information gained in Phase I will be used to develop the telephone-based, tailored, dyadic problem-solving intervention for rural HF dyads tested in Phase II.

Phase II (Arm II) will be guided by qualitative and quantitative inquiry and include a single-group, repeated measures design with time and dyad-member as within-subject factors. A sample size of 60 dyads (120 participants) is desired based on a power analysis for repeated measures ANOVA with 4 time points, alpha level of .05, a medium effect size (f = 0.25), and 80% power, plus oversampling for potential attrition (20%). Following verbal informed consent via telephone, all dyads will be screened for cognitive impairment using the Telephone Interview for Cognitive Status (TICS) prior to baseline data collection, which will include a Sociodemographic and Clinical Survey, the Self-Care of HF Index (SCHFI; v. 6.2) (patients only), the Caregiver Contribution to the Self-Care of HF Index (CCSCHFI) (caregivers only), Healthcare Utilization Survey, the Social Problem-Solving Inventory Revised-Short (SPSIRS), the Center for Epidemiological Studies-Depression (CESD), the Global Family Function Subscale (GFF) of the Family Assessment Device Questionnaire, and the Interpersonal Support Evaluation List-12 (ISEL-12). Caregivers will also complete the Dutch Objective Burden Inventory (DOBI), Denyes Self-care Practice Instrument (DENYES), and the BAKAS Caregiving Outcomes Scale (BAKAS).

Using a single group design, all dyads will participate in a problem-solving training intervention over 12 weeks (Weeks 1-4, 6, 8, 10, 12), with follow-up data collection occurring at weeks 5, 9, 11, 13. Qualitative data will be collected at weeks 5 and 11 via semi-structured interviews with dyads. Quantitative data on study outcomes and covariates will be collected at weeks 5, 9, and 13 and consist of the SCHFI (patient), CCSCHFI (caregiver), healthcare utilization (patient), SPSIRS (dyad), REALM (dyad), CESD (dyad), GFF (dyad),ISEL-12 (dyad), DOBI (caregiver), Denyes (caregiver) and the BAKAS (caregiver). All data will be self-report and collected by a trained research assistant who will collect study data over the telephone and mark participants answers on a computerized data spreadsheet. Qualitative data will be analyzed using thematic analytic methods and NVivo11. Possible treatment effectiveness on dyadic problem-solving, patient and caregiver contributions to HF self-care, healthcare utilization, caregiver burden, caregiver self-care, caregiver life changes, and differences among subgroups (gender, relationship type) over the 13 weeks will be examined using multilevel modeling and dyadic Growth Curve Modeling (GCM).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* consist of a patient with New York Heart Association Class II- IV HF and their family caregiver
* live in a rural area
* read, write, and communicate verbally in English
* have access to a telephone with speaker capability
* family caregivers are defined as a spouse/partner or adult family member living in the same household and/or considered to be the primary caregiver and may be healthy

Exclusion Criteria:

* patient has HF due to a correctable cause or condition
* either dyad member exhibits cognition dysfunction (i.e., score ≤ 30 on the Telephone Interview for Cognitive Status [TICS])

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-03-13 (Actual); Study Completion 2023-03-13 (Actual)

PRIMARY OUTCOMES:
Self-Care Maintenance (HF patient) | Baseline, 5 weeks
  Self-care maintenance will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Maintenance (HF patient) | Baseline, 9 weeks
  Self-care maintenance will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Maintenance (HF patient) | Baseline, 13 weeks
  Self-care maintenance will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to treatment adherence and self-monitoring. Scores are standardized (0-100), with higher scores suggesting better self-care maintenance. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Management (HF patient) | Baseline, 5 weeks
  Self-care management will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Management (HF patient) | Baseline, 9 weeks
  Self-care management will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Management (HF patient) | Baseline, 13 weeks
  Self-care management will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting better self-care management. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Confidence (HF patient) | Baseline, 5 weeks
  Self-care confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Confidence (HF patient) | Baseline, 9 weeks
  Self-care confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Self-Care Confidence (HF patient) | Baseline, 13 weeks
  Self-care confidence will be self-reported and measured using the Self-care of Heart Failure Index (SCHFI) v. 6.2. Items pertain to one's confidence in their ability to perform self-care activities. Scores are standardized (0-100), with higher scores suggesting better self-care confidence. Scores ≥ 70 are considered adequate, with an improvement of 8 or more considered clinically significant.
Caregiver Contribution to Self-Care Maintenance (caregiver) | Baseline, 5 weeks
  Caregiver contribution to self-care maintenance will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to treatment adherence and symptom monitoring. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care maintenance.
Caregiver Contribution to Self-Care Maintenance (caregiver) | Baseline, 9 weeks
  Caregiver contribution to self-care maintenance will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to treatment adherence and symptom monitoring. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care maintenance.
Caregiver Contribution to Self-Care Maintenance (caregiver) | Baseline, 13 weeks
  Caregiver contribution to self-care maintenance will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to treatment adherence and symptom monitoring. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care maintenance.
Caregiver Contribution to Self-Care Management (caregiver) | Baseline, 5 weeks
  Caregiver contribution to self-care management will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care management.
Caregiver Contribution to Self-Care Management (caregiver) | Baseline, 9 weeks
  Caregiver contribution to self-care management will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care management.
Caregiver Contribution to Self-Care Management (caregiver) | Baseline, 13 weeks
  Caregiver contribution to self-care management will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to symptom recognition and treatment and evaluation of treatment effectiveness. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care management.
Caregiver Contribution to Self-Care Confidence (caregiver) | Baseline, 5 weeks
  Caregiver contribution to self-care confidence will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to confidence in self-care ability. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care confidence.
Caregiver Contribution to Self-Care Confidence (caregiver) | Baseline, 9 weeks
  Caregiver contribution to self-care confidence will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to confidence in self-care ability. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care confidence.
Caregiver Contribution to Self-Care Confidence (caregiver) | Baseline, 13 weeks
  Caregiver contribution to self-care confidence will be self-reported and measured using the Caregiver Contribution to Self-care of Heart Failure Index (SCHFI). Items pertain to one's contribution to confidence in self-care ability. Scores are standardized (0-100), with higher scores suggesting higher contribution to self-care confidence.

SECONDARY OUTCOMES:
Healthcare Utilization (patient) | baseline, 5 weeks
  Healthcare utilization will be determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.
Healthcare Utilization (patient) | baseline, 9 weeks
  Healthcare utilization will be determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.
Healthcare Utilization (patient) | baseline, 13 weeks
  Healthcare utilization will be determined by the frequency of emergency department visits and 30-day readmissions for HF and assessed via self-report.
Problem-Solving (HF patient and caregiver) | baseline, 5 weeks
  Problem-solving will be self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving (HF patient and caregiver) | baseline, 9 weeks
  Problem-solving will be self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.
Problem-Solving (HF patient and caregiver) | baseline,13 weeks
  Problem-solving will be self-reported and assessed using the Social Problem-Solving Inventory Revised (SPSIR) which measures problem orientation and problem-solving style. In addition to a total score, there are 5 sub-scales: positive problem orientation, negative problem orientation, rational problem-solving, impulsivity/carelessness, and avoidance style. Higher scores on each sub-scale suggest more of the problem-solving characteristic. Higher total scores suggest more adaptive problem-solving, while lower scores indicate more maladaptive problem-solving.

OTHER OUTCOMES:
Depression (patient and caregiver) | baseline, 5 weeks
  Depression will be self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Depression (patient and caregiver) | baseline, 9 weeks
  Depression will be self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Depression (patient and caregiver) | baseline, 13 weeks
  Depression will be self-reported and assessed using the 20-item Center for Epidemiological Studies-Depression Scale (CES-D). The CES-D measures the presence of depression. Scores range from 0-60, with higher scores indicative of more symptoms of depression. A cut-off score ≥ 16 indicates depressed versus non-depressed.
Family Function (patient and caregiver) | baseline, 5 weeks
  Family function will be self-reported and measured using the Global Family Function (GFF) Subscale of the Family Assessment Device Questionnaire (12-items.The GFF assesses perception of overall family health related to problem-solving, communication, roles, active responses, affective involvement, and behavior control. Final mean scores range from 1 to 4 (healthy to unhealthy family functioning).
Family Function (patient and caregiver) | baseline, 9 weeks
  Family function will be self-reported and measured using the Global Family Function (GFF) Subscale of the Family Assessment Device Questionnaire (12-items.The GFF assesses perception of overall family health related to problem-solving, communication, roles, active responses, affective involvement, and behavior control. Final mean scores range from 1 to 4 (healthy to unhealthy family functioning).
Family Function (patient and caregiver) | baseline, 13 weeks
  Family function will be self-reported and measured using the Global Family Function (GFF) Subscale of the Family Assessment Device Questionnaire (12-items.The GFF assesses perception of overall family health related to problem-solving, communication, roles, active responses, affective involvement, and behavior control. Final mean scores range from 1 to 4 (healthy to unhealthy family functioning).
Social Support (patient and caregiver) | baseline, 5 weeks
  Social support will be self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.
Social Support (patient and caregiver) | baseline, 9 weeks
  Social support will be self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.
Social Support (patient and caregiver) | baseline, 13 weeks
  Social support will be self-reported and assessed using the Interpersonal Support and Evaluation List - 12 (ISEL-12) which measures perceived belonging, tangible, and appraisal support. Scores range from 0-36, with higher scores suggesting a higher perception of available support.
Caregiver Burden (caregiver) | baseline, 5 weeks
  Caregiver burden will be self-reported and assessed using the Dutch Objective Burden Inventory (DOBI), which measures both objective and subjective burden. Responses for each item range from 1 (no, never, not at all burdensome) to 3 (yes, often or always, very burdensome), with total scores on each subscale ranging from 1-3. Higher scores indicate greater perceived objective and subjective burden.
Caregiver Burden (caregiver) | baseline, 9 weeks
  Caregiver burden will be self-reported and assessed using the Dutch Objective Burden Inventory (DOBI), which measures both objective and subjective burden. Responses for each item range from 1 (no, never, not at all burdensome) to 3 (yes, often or always, very burdensome), with total scores on each subscale ranging from 1-3. Higher scores indicate greater perceived objective and subjective burden.
Caregiver Burden (caregiver) | baseline, 13 weeks
  Caregiver burden will be self-reported and assessed using the Dutch Objective Burden Inventory (DOBI), which measures both objective and subjective burden. Responses for each item range from 1 (no, never, not at all burdensome) to 3 (yes, often or always, very burdensome), with total scores on each subscale ranging from 1-3. Higher scores indicate greater perceived objective and subjective burden.
Caregiver Self-care (caregiver) | baseline, 5 weeks
  Caregiver self-care will be measured using the 18-item Denyes Self-care Practice Instrument (DENYES) which measures self-care activities that are universal self-care requisites (e.g., diet, rest, exercise, etc.). Response options for each item range from 0 to 156, with a total score calculated by averaging the time responses for all behaviors, with higher scores representing better self-care.
Caregiver Self-care (caregiver) | baseline, 9 weeks
  Caregiver self-care will be measured using the 18-item Denyes Self-care Practice Instrument (DENYES) which measures self-care activities that are universal self-care requisites (e.g., diet, rest, exercise, etc.). Response options for each item range from 0 to 156, with a total score calculated by averaging the time responses for all behaviors, with higher scores representing better self-care.
Caregiver Self-care (caregiver) | baseline, 13 weeks
  Caregiver self-care will be measured using the 18-item Denyes Self-care Practice Instrument (DENYES) which measures self-care activities that are universal self-care requisites (e.g., diet, rest, exercise, etc.). Response options for each item range from 0 to 156, with a total score calculated by averaging the time responses for all behaviors, with higher scores representing better self-care.
Life Changes (caregiver) | baseline, 5 weeks
  Caregiving-related life changes will be measured using the 15-item Bakas Caregiving Outcomes Scale. This instrument measures care partners' perceptions of how caregiving has influenced their social functioning, subjective well-being, and physical health using a 7-point (-3 [1] to +3 [7]) Likert-type scale. Total scores range from 15 to 105, with higher scores indicating more positive caregiving-related life changes.
Life Changes (caregiver) | baseline, 9 weeks
  Caregiving-related life changes will be measured using the 15-item Bakas Caregiving Outcomes Scale. This instrument measures care partners' perceptions of how caregiving has influenced their social functioning, subjective well-being, and physical health using a 7-point (-3 [1] to +3 [7]) Likert-type scale. Total scores range from 15 to 105, with higher scores indicating more positive caregiving-related life changes.
Life Changes (caregiver) | baseline, 13 weeks
  Caregiving-related life changes will be measured using the 15-item Bakas Caregiving Outcomes Scale. This instrument measures care partners' perceptions of how caregiving has influenced their social functioning, subjective well-being, and physical health using a 7-point (-3 [1] to +3 [7]) Likert-type scale. Total scores range from 15 to 105, with higher scores indicating more positive caregiving-related life changes.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Tallahassee Memorial Hospital Physician Partners - Blountstown Clinic, Blountstown, Florida
  - Tallahassee Memorial Hospital Physician Partners - Wakulla Clinic, Crawfordville, Florida
  - Talllahassee Memorial Physician Partners Cardiology - Marianna Clinic, Marianna, Florida
  - Tallahassee Memorial Hospital Physician Partners - Monticello Clinic, Monticello, Florida
  - Tallahassee Memorial Hospital Physician Partners - Perry Clinic, Perry, Florida
  - Tallahassee Memorial Hospital Physician Partners - Quincy Clinic, Quincy, Florida
  - Bond Community Health Center, Tallahassee, Florida
  - Tallahassee Memorial Hospital Physician Partners Cardiology Heart Failure Clinic, Tallahassee, Florida
  - HCA Capital Cardiology Associates, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers.